CLINICAL TRIAL: NCT03369925
Title: A Parallel, Double-Blind Study to Assess the Cognitive Effects of a Citicoline Supplement (Cognizin®) in Men and Women With Age-Associated Memory Impairment
Brief Title: Cognitive Effects of Citicoline in Men and Women With Age-Associated Memory Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyowa Hakko Bio Co., Ltd. (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BIO-1707
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo supplement
- Cognizin (Experimental)
  Interventions: Dietary Supplement: Citicoline supplement

INTERVENTIONS:
Dietary Supplement: Placebo supplement — Cellulose
  Other Names: Placebo
  Arms: Placebo
Dietary Supplement: Citicoline supplement — Cognizin
  Other Names: Cognizin
  Arms: Cognizin

SUMMARY:
The objective of this trial is to determine the effects of citicoline on cognitive performance in healthy Men and Women with Age-Associated Memory Impairment compared to a placebo.

DETAILED DESCRIPTION:
This study is a 12-week, randomized, double-blind, placebo-controlled trial of citicoline in healthy men and women with Age-Associated Memory Impairment. Cognitive assessments will be performed to determine whether citicoline administration with supportive memory, compared to placebo administration.

ELIGIBILITY:
Inclusion Criteria:

* male or female, 50-85 years of age
* at least a high school diploma or the equivalent
* self-reported memory loss
* scores ≥24 on the Mini-Mental State Examination, ≥85 on the Kaufman Brief Intelligence Test, Second Edition, ≤5 on the Geriatric Depression Scale, and 4, 3, or 2 on the Spatial Span Test
* no health conditions that would prevent him or her from fulfilling the study requirements on the basis of medical history and routine laboratory test results

Exclusion Criteria:

* color blind
* abnormal laboratory test results
* major medical or neurological illness
* female who is pregnant, planning to be pregnant during the study period
* requiring treatment with a drug which might obscure the action of the study treatment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Standardized scores on the Cambridge Brain Sciences that measure cognitive assessment | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Clinical Research, Inc., Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nakazaki E, Mah E, Sanoshy K, Citrolo D, Watanabe F. Citicoline and Memory Function in Healthy Older Adults: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. J Nutr. 2021 Aug 7;151(8):2153-2160. doi: 10.1093/jn/nxab119. PMID 33978188